CLINICAL TRIAL: NCT04418167
Title: A Phase 1 Study of ERK1/2 Inhibitor JSI-1187 Administered as Monotherapy and in Combination With Dabrafenib for the Treatment of Advanced Solid Tumors With MAPK Pathway Mutations
Brief Title: JSI-1187-01 Monotherapy and in Combination With Dabrafenib for Advanced Solid Tumors With MAPK Pathway Mutations
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: JS InnoPharm, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JSI-1187-01
Record Dates: First submitted 2020-05-11; First posted 2020-06-05 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors
Keywords: solid tumor; neoplasm; BRAF V600 mutation; MAPK pathway mutation; ERK1/2; JSI-1187; Dabrafenib; KRAS; NRAS; BRAF; melanoma; non-small cell lung cancer; anaplastic thyroid cancer
MeSH Terms: conditions — Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Thyroid Carcinoma, Anaplastic | interventions — dabrafenib

STUDY DESIGN:
Intervention Model Description: A total of up to 80 subjects are anticipated in the JSI-1187 monotherapy dose-escalation phase (Part A). A total of up to 36 subjects are anticipated in the JSI-1187 plus dabrafenib dose-escalation phase (Part B). A total of 58 subjects are anticipated in the JSI-1187 plus dabrafenib expansion phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: JSI-1187 Monotherapy Dose Escalation (Experimental): Locally advanced or metastatic solid tumors with confirmed with MAPK pathway mutation
  Interventions: Drug: JSI-1187
- Part B: JSI-1187 Plus Dabrafenib Combination Dose Escalation (Experimental): BRAF V600E/K-mutated unresectable or metastatic melanoma, BRAF V600E-mutated NSCLC, or BRAF V600E-mutated locally advanced or metastatic anaplastic thyroid cancer, or other BRAF V600E-mutated unresectable or metastatic solid tumors
  Interventions: Drug: JSI-1187; Drug: Dabrafenib
- Part C: JSI-1187 Plus Dabrafenib Expansion (Experimental): Cohort 1: BRAF V600E/K-mutated unresectable or metastatic melanoma after 1-3 prior therapies for metastatic disease, including anti-PD1 therapy, with or without ipilimumab, and BRAF/MEK inhibitor treatment.
  Cohort 2: BRAF V600E/K-mutated unresectable or metastatic melanoma after BRAF/MEK inhibitor adjuvant therapy for Stage 3 disease followed by 1-2 prior therapies for metastatic disease, including anti-PD-1 therapy, with or without ipilimumab, and excluding BRAF/MEK inhibitor treatment.
  Cohort 3: BRAF V600E-mutated metastatic NSCLC after 1-2 prior therapies for metastatic disease.
  Interventions: Drug: JSI-1187; Drug: Dabrafenib

INTERVENTIONS:
Drug: JSI-1187 — JSI-1187 capsules for oral administration
Drug: Dabrafenib — Dabrafenib capsules for oral administration
  Other Names: TAFINLAR
  Arms: Part B: JSI-1187 Plus Dabrafenib Combination Dose Escalation; Part C: JSI-1187 Plus Dabrafenib Expansion

SUMMARY:
This is a Phase 1 study of JSI-1187 as monotherapy and in combination with dabrafenib for the treatment of advanced solid tumors with MAPK pathway mutations, including mutations that cause MAPK pathway hyperactivation.

DETAILED DESCRIPTION:
Selected subjects will include males and females age ≥18 years; histologically confirmed locally advanced or metastatic solid tumors with archived tumor sample from the primary, recurrent or metastatic disease with documented MAPK pathway mutation or pathway hyperactivating mutations; advanced or recovered from all acute toxicities (≤ Grade 1) due to prior therapy; adequate renal and hepatic function; and no known history of significant cardiac or retinal disease.

Part A (Monotherapy Dose Escalation): Following screening, a total of up to 80 subjects are anticipated to establish the MTD of JSI-1187 monotherapy in subjects with locally advanced or metastatic solid tumors with MAPK pathway mutations, including hyperactivating pathway mutations or gene fusions, refractory to or relapsed on prior therapy. JSI-1187 will be administered orally at doses of 2, 4 and 8 mg twice daily, and at doses of 16, 24, 36, 56, 88 and 128 mg once or twice daily, or until an MTD for both regimens is reached, whichever is earlier, repeated every 28 days (=1 cycle). A 3+3 dose escalation schema will be followed to establish the MTD of the JSI-1187 monotherapy. Subjects will take their doses in a fasted state, 1 hour before or 2 hours after a meal. A total of 6 subjects will be treatment at the MTD before starting Part B.

(On hold, effective 05 July 2023) Part B (Combination Dose Escalation): Following screening, a total of up to 36 subjects are anticipated to establish the MTD of JSI-1187 plus dabrafenib in BRAF V600E/K-mutated unresectable or metastatic melanoma, BRAF V600E-mutated metastatic non-small cell lung cancer (NSCLC), BRAF V600E-mutated locally advanced or metastatic anaplastic thyroid cancer, or other BRAF V600E-mutated unresectable or metastatic solid tumors. A 3+3 dose escalation schema will be followed to establish the MTD of the JSI-1187 plus dabrafenib combination. Daily doses of both drugs will be taken in the fasted state. A total of 6 subjects will be treated at the JSI-1187 plus dabrafenib combined MTD before beginning Part C.

(On hold, effective 05 July 2023) Part C (Expansion Cohorts): Following screening, a total of 58 subjects in 3 cohorts are anticipated to expand the disease treatment settings of JSI-1187 in combination with dabrafenib in BRAF V600E/K-mutated melanoma or BRAF V600E-mutated NSCLC.

Cohort 1: JSI-1187 plus dabrafenib in BRAF V600E/K-mutated unresectable or metastatic melanoma after 1-3 prior therapies for metastatic disease, including anti-PD1 therapy, with or without ipilimumab, and BRAF/MEK inhibitor treatment. (n=21).

Cohort 2: JSI-1187 plus dabrafenib in BRAF V600E/K-mutated unresectable or metastatic melanoma after BRAF/MEK inhibitor adjuvant therapy for Stage 3 disease followed by 1-2 prior therapies for metastatic disease, including anti-PD-1 therapy, with or without ipilimumab, and excluding BRAF/MEK inhibitor treatment. (n=21).

Cohort 3: JSI-1187 plus dabrafenib in BRAF V600E-mutated metastatic NSCLC after 1-2 prior therapies for metastatic disease. (n=16).

JSI-1187 plus dabrafenib will be administered at the MTDs established for both drugs in Part B, repeated every 28 days (=1 cycle).

Subjects who demonstrate clinical benefit (CR, PR or SD) will be allowed to continue therapy with JSI-1187 (and dabrafenib) until progression of disease, observation of unacceptable adverse events, intercurrent illness or changes in the subject's condition that prevents further study participation.

Disease response will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST v.1.1).

Blood for hematology, coagulation parameters and serum chemistry determinations will be collected, ECGs will be taken, and ophthalmologic exams will be conducted during the study.

Blood will be collected for PK assessment of JSI-1187 and PD assessment of pRSK/RSK ratio determinations.

Tumor biopsies (optional) will be collected from consenting subjects at Screening and on-study for pRSK determination. Results will be correlated with clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* Have locally advanced or metastatic solid tumor malignancy with measurable disease and be an appropriate candidate for experimental therapy
* Part A (JSI-1187 Monotherapy Dose Escalation): Histologically or cytologically confirmed MAPK pathway mutation, including hyperactivating pathway mutations or gene fusions, e.g., BRAF (Class I, II or III), RAS (H/K/N), MEK (MAP2K1), RAS-GAP (NF1 loss, RASA1), RAS-GEF, refractory to or relapsed on prior therapy, and have received all available therapy known to confer clinical benefit
* (On hold, effective 05 July 2023) Part B (JSI-1187 Plus Dabrafenib Combination Dose Escalation): Histologically or cytologically confirmed BRAF V600E/K-mutated unresectable or metastatic melanoma, BRAF V600E-mutated metastatic NSCLC, BRAF V600E-mutated locally advanced or metastatic anaplastic thyroid cancer, or other BRAF V600E-mutated unresectable or metastatic solid tumors, refractory to, or relapsed on, prior therapy, and have received all available therapy known to confer clinical benefit
* (On hold, effective 05 July 2023) Part C (JSI-1187 Plus Dabrafenib Expansion Cohorts): Histologically or cytologically confirmed:

  * Cohort 1: BRAF V600E/K-mutated unresectable or metastatic melanoma after 1-3 prior therapies for metastatic disease, including anti-PD1 therapy, with or without ipilimumab, and BRAF/MEK inhibitor treatment
  * Cohort 2: BRAF V600E/K-mutated unresectable or metastatic melanoma after BRAF/MEK inhibitor adjuvant therapy for Stage 3 disease followed by 1-2 prior therapies for metastatic disease, including anti-PD-1 therapy, with or without ipilimumab, and excluding BRAF/MEK inhibitor treatment
  * Cohort 3: BRAF V600E-mutated metastatic NSCLC after 1 or 2 prior therapies for metastatic disease
* MAPK mutation tumor status will be established prior to entry based on previous MAPK pathway mutation reports from a CLIA qualified laboratory, or, if a report is not available, the mutation analysis will be performed at Screening on archival tissue or newly biopsied tumor tissue.
* Have discontinued previous treatments for cancer and have resolution, except where otherwise stated in the inclusion criteria, of all clinically significant toxic effects of prior cancer treatment, surgery, or radiotherapy to Grade ≤ 1. Subjects with prior immune checkpoint inhibitor endocrinopathies must have resolution to ≤ Grade 2 and be stable on hormonal therapy (e.g., levothyroxine, hydrocortisone, insulin, etc.).
* Adequate performance status: Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy of ≥ 3 months
* Subjects with asymptomatic stable, prior or currently treated brain metastases are allowed
* Adequate hematologic parameters without ongoing transfusional support:

  * Hemoglobin (Hb) ≥ 9 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9 cells/L
  * Platelets ≥ 75 x 10^9 cells/L
* Adequate renal and hepatic function:

  * Creatinine ≤ 1.5 times the upper limit of normal (ULN), or calculated creatinine clearance ≥ 50 mL/minute x 1.73 m^2 per the Cockcroft-Gault formula
  * Total bilirubin ≤ 1.5 times the (ULN) unless due to Gilbert's disease
  * ALT/AST ≤ 2 times the ULN, or < 3 times the ULN for subjects with liver metastases
* Negative serum pregnancy test within 14 days prior to the first dose of study therapy for women of child-bearing potential (WCBP). Sexually active WCBP and male subjects must agree to use adequate methods to avoid pregnancy throughout the study and for 28 days after the completion of study treatment.
* Ability to provide written informed consent

Exclusion Criteria:

* Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV
* QT interval corrected for rate (QTc) > 480 msec on the ECG obtained at Screening using Fridericia method for QTc calculation
* Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes, with the exception of anti-microbials that are used as standard of care to prevent or treat infections and other such drugs that are considered by the Investigator to be essential for patient care.
* Medications that are strong inhibitors of CYP3A4 are prohibited during study and for 14 days prior to the first dose of study drug(s).
* Medications that are strong inducers of CYP3A4 are prohibited during study and for 14 days prior to the first dose of study drug(s).
* Medications that are strong inhibitors of BCRP are prohibited during study and for 14 days prior to the first dose of study drugs(s).
* Subjects on dabrafenib (Parts B and C) also are advised to avoid concurrent administration of strong inhibitors of CYP2C8 as these medications may increase the concentration of dabrafenib
* History of or current evidence/risk of retinal vein occlusion or central serous retinopathy, or has medically relevant abnormalities identified on screening ophthalmologic examination
* Symptomatic central nervous system malignancy or metastasis
* Gastrointestinal conditions that could impair absorption of study drug(s)
* Current hematologic malignancies
* Second, active primary solid tumor malignancy that, in the judgement of the investigator or Sponsor medical monitor, may affect the interpretation of results
* Prior malignancies, with the exception of carcinoma in situ of any origin, non-muscle invasive bladder cancer, Gleason 3+3 prostate cancer and prior malignancies in remission whose likelihood of recurrence is very low, as judged by the Sponsor medical monitor.
* Active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) requiring treatment within the last week prior to study treatment
* Other active infection requiring IV antibiotic usage within the last week prior to study treatment
* Any other medical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results
* Receipt of an investigational product on a clinical trial within 5 elimination half-lives or within 28 days, whichever is shorter, prior to C1D1 on this study, or currently enrolled in a clinical trial, involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Previously completed or withdrawn from this study or any other study investigating an ERK1/2 inhibitor.
* If female, pregnant, breast-feeding, or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (safety and tolerability) | 35 months
  Safety and tolerability assessed by adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Objective Response Rate | Assessed at the end of Cycle 2 and every 2 cycles thereafter through 6 months following last dose of study drug (each cycle is 28 days)
  Proportion of subjects with objective responses (complete response [CR] + partial response [PR]) as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1.
Duration of Response | Assessed at the end of Cycle 2 and every 2 cycles thereafter through 6 months following the last dose of study drug (each cycle is 28 days)
  Length of time from first evidence of objective response (CR, PR) to the first objective evidence of disease progression
Time to Response | Assessed at the end of Cycle 2 and every 2 cycles thereafter through 6 months following the last dose of study drug (each cycle is 28 days)
  Length of time from the date of first dose of study drug to the first evidence of objective response (CR, PR)
Disease Control Rate | Assessed at the end of Cycle 2 and every 2 cycles thereafter through 6 months following the last dose of study drug (each cycle is 28 days)
  Proportion of subjects with best response of CR, PR or stable disease (SD)
Progression-Free Survival | Assessed from the date of the first dose of study drug to the first evidence of disease progression or death, whichever is earlier, assessed up to 35 months
  Length of time from the date of first dose of study drug to the first evidence of disease progression or death, whichever is earlier
Overall Survival | Assessed from the date of the first dose of study drug to date of death from any cause, assessed up to 35 months
  Length of time from the date of first dose of study drug to date of death from any cause

OTHER OUTCOMES:
Mean plasma concentrations of JSI-1187 alone and in combination with dabrafenib | Cycle 1, Day 1; Cycle 1, Day 15; Cycle 2 Day 1; Cycle 4 Day 1; Cycle 6 Day 1 (each cycle is 28 days)
  Mean plasma concentrations of JSI-1187 will be determined as monotherapy, and when given in combination with dabrafenib, and summarized by dose group.
pRSK/RSK ratio in whole blood (PBMCs) (pharmacodynamic endpoint) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
  Change from baseline in whole blood (PBMC) pRSK/RSK ratio will be determined and summarized by dose group.
Change in pRSK levels in tumor (pharmacodynamic endpoint) | At Screening and Week 2 or 3 on study
  In consenting subjects and when clinically available, tumor biopsies will be taken pre-study and on study to assess change in tumor pRSK.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - University of Arizona Comprehensive Cancer Center, Tucson, Arizona
  - University of California Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No